CLINICAL TRIAL: NCT05927597
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses and the Open-Label Food Effect of a Single Dose of INS1007 in Healthy Japanese and Caucasian Subjects
Brief Title: A Study of the Safety, Pharmacokinetics, and Pharmacodynamics of INS1007 in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1007-101
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Cohort 1 (Dose 1) (Experimental): Japanese and Caucasian participants will receive INS1007 at Dose 1 or matching placebo, orally, once on Day 1, and Day 4 through Day 30 in Part A under fasted conditions.
  Interventions: Drug: INS1007; Drug: Placebo
- Part A: Cohort 2 (Dose 2) (Experimental): Japanese and Caucasian participants will receive INS1007 at Dose 2 or matching placebo, orally, once on Day 1, and Day 4 through Day 30 in Part A under fasted conditions.
  Interventions: Drug: INS1007; Drug: Placebo
- Part A: Cohort 3 (Dose 3) (Experimental): Japanese and Caucasian participants will receive INS1007 at Dose 3 or matching placebo, orally, up to Day 30 in Part A under fasted conditions. Enrollment will commence in this cohort once the safety and tolerability data in Cohort 2 is deemed acceptable by the principal investigator (PI) and the Sponsor's medical monitor.
  Interventions: Drug: INS1007; Drug: Placebo
- Part B: Treatment Sequence 1 (Experimental): Japanese and Caucasian participants will receive INS1007 at the dose established in Part A after a high-fat and high-calorie breakfast on Day 1 followed by a dose established in Part A on Day 8 under fasted conditions in Part B of the study.
  Interventions: Drug: INS1007
- Part B: Treatment Sequence 2 (Experimental): Japanese and Caucasian participants will receive INS1007 at the dose established in Part A under fasted conditions on Day 1 followed by dose established in Part A on Day 8 after a high-fat and high-calorie breakfast in Part B of the study.
  Interventions: Drug: INS1007

INTERVENTIONS:
Drug: INS1007 — Oral tablets.
  Other Names: AZD7986; Brensocatib
Drug: Placebo — Oral tablets.
  Arms: Part A: Cohort 1 (Dose 1); Part A: Cohort 2 (Dose 2); Part A: Cohort 3 (Dose 3)

SUMMARY:
The primary purpose of Part A of this study is to compare, in a single dose and multiple doses the safety, tolerability, and pharmacokinetics (PK) profile administered in Japanese and Caucasian participants and of Part B of the study is to assess the food effect of a single dose of INS1007 administered in Japanese and Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

* For Japanese participants: Participant is of Japanese descent as evidenced by verbal confirmation of familial heritage (a participant must have all four grandparents born in Japan). Participants must have lived less than 10 years outside of Japan.
* For Caucasian participants: Participants must be of Caucasian descent, as evidenced by verbal confirmation that all four grandparents are Caucasian.
* Healthy, based on pre-study medical evaluation (medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations) by the PI or designee.

Exclusion Criteria:

* Have clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the PI or designee.
* Have had serious, opportunistic, or chronic/recurring infection within 6 months prior to Screening. Examples may include, but are not limited to, infections requiring intravenous (IV) antibiotics, hospitalization, or prolonged (>14 day) anti-infective treatment.
* Have a history of multiple or severe allergies, or an anaphylactic reaction, to prescription or non-prescription drugs or food.
* Have a positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody, or human immunodeficiency virus (HIV) antigen or antibody at the Screening Visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Number of Participants Who Experienced at Least One Adverse Event (AE) | Up to Day 61 in Part A and up to Day 11 in Part B
  Determination and comparison of the safety and tolerability of INS1007 following single and multiple dose administration in Japanese and Caucasian participants.
Parts A and B: Area Under the Plasma Concentration-time Curve (AUC) of INS1007 | Part A: Predose and at multiple time points postdose up to Day 33; Part B: Predose and at multiple time points postdose up to Day 11
  Comparison of the pharmacokinetics of single and multiple doses of INS1007 in Japanese and Caucasian participants.

SECONDARY OUTCOMES:
Part A: Pharmacodynamic Activity Based on Concentration of Biomarkers in Blood | Up to Day 61
  Pharmacodynamic activity based on concentration of biomarkers cathepsin G (Cat G), proteinase 3 (PR3), neutrophil elastase (NE), and absolute neutrophil in blood will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Usansky H, Yoon E, Teper A, Zou J, Fernandez C. Safety, Tolerability, and Pharmacokinetic Evaluation of Single and Multiple Doses of the Dipeptidyl Peptidase 1 Inhibitor Brensocatib in Healthy Japanese and White Adults. Clin Pharmacol Drug Dev. 2022 Jul;11(7):832-842. doi: 10.1002/cpdd.1094. Epub 2022 Apr 11. PMID 35411669
- See also: Results are available in the link to the publication. — https://pubmed.ncbi.nlm.nih.gov/35411669/